CLINICAL TRIAL: NCT06376357
Title: Roles in the Management of Treatment-Induced Peripheral Neuropathy in Cancer Patients Receiving Taxane-Based Chemotherapy and the Effect of Foot Massage on Neuropathy and Quality of Life: A Randomized Controlled Study
Brief Title: The Effect of Foot Massage With Roles on Cancer Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ülkü Saygılı, Assist. Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16.04.24/1
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Neoplasms; Over Cancer; Foot Massage
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental)
  Interventions: Other: Foot Massage with roller
- Control (No Intervention)

INTERVENTIONS:
Other: Foot Massage with roller — The intervention group is expected to apply roller massage to the soles of both feet in a sitting position on a chair (8 hours apart at 08.00, 16.00, 24.00 hours) every day for 6 weeks, 3x5 minutes a day. Video recording will be used as a reminder in the application.
  Arms: Study

SUMMARY:
It was aimed to examine the roles in the management of treatment-related peripheral neuropathy in cancer patients receiving taxane-based chemotherapy and the effect of foot massage on neuropathy and quality of life.

DETAILED DESCRIPTION:
Intervention Phase of the Research;

1. Patient information about neuropathy caused by chemotherapy and its management,
2. Teaching the role application to the patient,
3. Application process
4. It will be carried out in 4 steps, including patient monitoring via telemonitoring.

ELIGIBILITY:
Inclusion Criteria:

* Being registered in the medical oncology outpatient clinic of Selçuk University Faculty of Medicine Hospital
* Completed standard taxane-based chemotherapy treatment protocol for breast and ovarian cancer
* Karnofsky Performance Scale being 80 and above (Performance scale of cancer patients)
* Being 18 years or older
* Having received at least 3 cycles of taxane-based treatment
* Presence of grade 2 or higher peripheral neuropathy
* Being conscious and cooperative
* Verbal and written approval to participate in the study after an explanation about the study is made.

Exclusion Criteria:

* Previous skin sensitivity on hands and feet
* Refused to participate in the study after making a statement about the study
* Development of peripheral neuropathy due to reasons other than chemotherapy [tumor compression, nutritional disorders, infections or major systemic disease (diabetes mellitus, etc.)]
* Bone, spine metastasis or malignancy
* Having mental and psychic problems that would prevent him from taking part in the research.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-27 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ C-30 Quality of Life Scale | 10 minutes
  Quality of life of patients will be evaluated with EORTC QLQ-C30, which was developed by EORTC for cancer patients and is widely used all over the world.
CIPN20 Neuropathy Scale | 10 minutes
  It is a 20-item assessment tool used to reveal the symptoms of chemotherapy-related peripheral neuropathy and the impact of functional limitations caused by this problem on patients' lives.
One Leg Standing Test | 5 minutes
  The Single Leg Standing Test (TAUDT), which is widely used to evaluate static balance, is a simple test that can be used in many situations and requires minimal equipment.
Brief Pain Inventory BPI | 5 minutes
  The BPI questionnaire is a short, easy-to-apply assessment method that can be used to evaluate pain and related functions (general activity, walking ability, normal work, relationships with other people, sleep, enjoyment of life). It includes simple 0 to 10 numerical rating scales that are both easy to understand and easy to translate into different languages. In the short pain inventory, the mildest pain score = 0 and the most severe pain score = 10.
Pain Threshold Assessment Test | 5 minutes
  algometer (Baseline, USA) will be used. The Algometer (Relevant material is located in Selçuk University SHMYO application laboratory and it is planned to be taken and used with a report for the study and returned after the last measurements) is positioned upright and the pressure is increased to 1kg/cm2 at the painful point every three seconds and the measurements are taken with a 30-second rest period in between. It is applied 3 times and the average of 3 measurements is used for analysis.
Two Point Discrimination | 10 minutes
  Evaluation will be made from the trans-metatarsal area, middle of the foot and middle of the heel. It will start from the interval where two points can be easily distinguished. The distance between two points will be reduced in 1 mm intervals until the two points are felt as a single point. Then, it will start with two-point stimulation at the minimum interval felt as a single point, and the distance between the two points will be increased in 1 mm intervals until the distance between the two points is felt separately as two points again.

CONTACTS AND LOCATIONS:
Locations (1):
- ülkü Saygili Düzova, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No